CLINICAL TRIAL: NCT00036894
Title: A Phase I Trial Of A Thalidomide Analog, CC-5013, For The Treatment Of Patients With Recurrent High-Grade Gliomas
Brief Title: CC-5013 in Treating Patients With Recurrent Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069338; NCI-02-C-0145; NCT00032214 (obsolete NCT alias)
Record Dates: First submitted 2002-05-13; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2003-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult ependymoblastoma; adult anaplastic ependymoma; adult myxopapillary ependymoma; adult meningioma; adult meningeal hemangiopericytoma; adult brain stem glioma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Neuroectodermal Tumors, Primitive; Ependymoma; Meningioma; Gliosarcoma | interventions — Lenalidomide

INTERVENTIONS:
Drug: lenalidomide

SUMMARY:
RATIONALE: CC-5013 may stop the growth of gliomas by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of CC-5013 in treating patients who have recurrent glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of CC-5013 in patients with recurrent high-grade gliomas.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine the antiangiogenic activity of this drug in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to concurrent enzyme-inducing antiepileptic drugs (yes vs no).

Patients receive oral CC-5013 weekly for 3 weeks. Treatment repeats every 4 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CC-5013 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 2 weeks.

PROJECTED ACCRUAL: A maximum of 80 patients (40 per stratum) will be accrued for this study within 20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following:

  * Histologically confirmed high-grade glioma

    * Glioblastoma multiforme
    * Gliosarcoma
    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Anaplastic mixed oligoastrocytoma
    * Malignant glioma/astrocytoma, not otherwise specified
    * Meningioma
    * Hemangioblastoma
    * Ependymoma
    * Primitive neuroectodermal tumors
    * Hemangiopericytoma
    * Progressive glioma
  * Clinically and radiographically diagnosed brain stem glioma
* Progressive or recurrent disease as determined by CT scan or MRI

  * Biopsy allowed for prior recent (i.e., within the past 12 weeks) resection of recurrent or progressive tumor
* Must have failed prior radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 8 weeks

Hematopoietic:

* WBC at least 2,300/mm^3
* Platelet count at least 90,000/mm^3
* Hemoglobin at least 8 g/dL (transfusions allowed)

Hepatic:

* Bilirubin less than 3 times upper limit of normal (ULN)
* SGOT less than 3 times ULN
* No significant active hepatic disease

Renal:

* Creatinine less than 2.0 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No significant active renal disease

Cardiovascular:

* No significant active cardiac disease

Other:

* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No significant active psychiatric disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 2 weeks since prior interferon
* No concurrent immunotherapy

Chemotherapy:

* At least 6 weeks since prior nitrosoureas
* At least 4 weeks since prior temozolomide or carboplatin
* At least 3 weeks since prior procarbazine
* At least 2 weeks since prior vincristine
* At least 4 weeks since other prior cytotoxic chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* At least 2 weeks since prior tamoxifen
* Concurrent steroids allowed for control of the signs and symptoms of increased intracranial pressure if on a stable dose for at least the past 5 days

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 2 weeks since prior tumor resection

Other:

* At least 2 weeks since other prior noncytotoxic agents
* Concurrent enzyme-inducing antiepileptic drugs allowed
* No concurrent rifampin
* No concurrent grapefruit juice
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Fine, MD, Study Chair — NCI - Neuro-Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Fine HA, Kim L, Albert PS, Duic JP, Ma H, Zhang W, Tohnya T, Figg WD, Royce C. A phase I trial of lenalidomide in patients with recurrent primary central nervous system tumors. Clin Cancer Res. 2007 Dec 1;13(23):7101-6. doi: 10.1158/1078-0432.CCR-07-1546. PMID 18056189